CLINICAL TRIAL: NCT05958160
Title: Modified Atkins Diet Versus Topiramate In Children With Epileptic Spasms Refractory To Hormonal Treatment: A Randomized Open-Label Study
Acronym: TOPAMAD
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, Suvasini Sharma, Professor, Lady Hardinge Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOPAMAD
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Epileptic Spasms, Failed Hormonal Therapy
MeSH Terms: conditions — Spasms, Infantile | interventions — Diet, Ketogenic; Topiramate

STUDY DESIGN:
Intervention Model Description: Randomized Open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Atkins Diet Arm (Experimental): Modified Atkins diet will be added to the ongoing anti-seizure medication regimen
  Interventions: Other: Modified Atkins diet
- Topiramate arm (Active Comparator): Topiramate will be added to the ongoing anti-seizure medication regimen
  Interventions: Drug: Topiramate

INTERVENTIONS:
Other: Modified Atkins diet — The modified Atkins diet is a less restrictive version of the ketogenic diet
  Other Names: Ketogenic diet
  Arms: Modified Atkins Diet Arm
Drug: Topiramate — Topiramate is an anti-seizure medication
  Arms: Topiramate arm

SUMMARY:
This study has been planned to compare the efficacy and tolerability of topiramate, a commonly used second line agent, with modified Atkins diet in children with epileptic spasms refractory to hormonal treatment, in a randomized open label study.

DETAILED DESCRIPTION:
Infantile epileptic spasms syndrome, formerly known as West syndrome is a severe and difficult to treat epilepsy syndrome in infants and young children. The first-line options of this condition include hormonal therapy, i.e., adrenocorticotropic hormone (ACTH) or oral corticosteroids, and/or vigabatrin. These are effective in 45%-55% of the patients. These are however associated with significant side effects, and high relapse rates. Newer drugs such as topiramate, zonisamide, and levetiracetam have also been evaluated; but there have been no randomized trials to evaluate the efficacy of these agents. Topiramate is one of the most commonly used second line agents used for the treatment of epileptic spasms.

The ketogenic diet (KD), a high-fat, low-carbohydrate, adequate-protein diet is an established, effective non-pharmacologic treatment for children with intractable epilepsy. Despite being highly efficacious, ketogenic diet has practical constraints in implementation leading to need for alternative approaches. The modified Atkins diet is a less restrictive variation of the ketogenic diet. This diet is more palatable and acceptable in comparison to ketogenic diet. The modified Atkins diet has shown to be effective in children with epileptic spasms refractory to first line treatment in a recent randomized controlled trial, comparing add-on diet versus continuing the on-going anti-seizure medications alone. At the end of 4 weeks, 11 children in the diet group were spasm free compared with none in the control group (P ≤ .001).

This study has been planned to compare the efficacy and tolerability of topiramate, a commonly used second line agent, with modified Atkins diet in children with epileptic spasms refractory to hormonal treatment, in a randomized open label study. The results will guide clinicians as to the best options in children with epileptic spasms refractory to hormonal treatment.

ELIGIBILITY:
Inclusion Criteria:

1) Age: 9 months to 3 years 2) Diagnosis of infantile epileptic spasms syndrome as per the ILAE 2022 diagnostic criteria 3) Failure of hormonal therapy, i.e. oral prednisolone or ACTH

-

Exclusion Criteria:

1) Known or suspected inborn error of metabolism 2) Prior use of the ketogenic or modified Atkins diet or Topiramate 3) Systemic illness- chronic hepatic, renal or pulmonary disease 4) Diagnosed renal stones

-

Ages: 9 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2023-07-20 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of children with ≥ 50% reduction in clinical spasms at 12 weeks as compared to baseline as per parental reports in both groups | 12 weeks
  The proportion of children with ≥ 50% reduction in clinical spasms at 12 weeks as compared to baseline as per parental reports in both groups

SECONDARY OUTCOMES:
The proportion of children with clinical spasm cessation as per parental reports at the end of 12 weeks of treatment in both groups. | 12 weeks
The proportion of children with ≥ 1 point improvement in BASED score at 12 week as compared to baseline in both groups | 12 weeks
Adverse effects of the intervention in both groups | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Suvasini Sharma, MD, DM, Principal Investigator — Lady Hardinge Medical College
Locations (1):
- Lady Hardinge Medical College and Associated Kalawati Saran Children's Hospital, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Meena R, Roy Chowdhury S, Elwadhi A, Jain P, Mukherjee SB, Sharma S. Modified Atkins diet versus topiramate in young children with epileptic spasms refractory to steroids and vigabatrin: a randomised open-label trial. Seizure. 2025 Sep;131:405-412. doi: 10.1016/j.seizure.2025.08.011. Epub 2025 Aug 10. PMID 40840039